CLINICAL TRIAL: NCT03262025
Title: Primary Cecal Pathologies Presenting as Acute Abdomen and Critical Appraisal of Their Current Management Strategies
Brief Title: Primary Cecal Pathologies Presenting as Acute Abdomen
Status: Completed | Type: Observational
Sponsor: Jawaharlal Nehru Medical College (Other)
Responsible Party: Principal Investigator, Kaushal Deep Singh, Principal Investigator, Jawaharlal Nehru Medical College
Other Study IDs: CecalJNMC
Record Dates: First submitted 2017-08-23; First posted 2017-08-25 (Actual); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Acute Abdomen; Emergency Surgery; Laparotomy; Amoebic Colitis; Diverticulitis of Caecum; Typhlitis
Keywords: Primary cecal pathology; Emergency laparotomy; Ruptured liver abscess; Right hemicolectomy; Conservative colonic resection; Fulminant amoebic colitis; Ileocecal resection; Ileoascending anastomosis; Ileotransverse anastomosis; Cecal diverticulitis; Amoebic typhilitis; Idiopathic typhilitis
MeSH Terms: conditions — Abdomen, Acute; Dysentery, Amebic; Typhlitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Operated patients who survived: Patients who were discharged in index hospital admission after operative intervention
  Interventions: Procedure: Operated
- Operated patients who expired: Patients who expired in index hospital admission after operative intervention
  Interventions: Procedure: Operated
- Non-operated patients who survived: Patients who were discharged in index hospital admission after being managed conservatively
- Non-operated patients who expired: Patients who expired in index hospital admission after being managed conservatively

INTERVENTIONS:
Procedure: Operated — Patients were either managed conservatively or underwent emergency laparotomy
  Groups: Operated patients who expired; Operated patients who survived

SUMMARY:
Background: The importance of cecal pathologies lie in the fact that being the first part of large intestine, any disease involving the cecum affects overall functioning of the large bowel. Primary cecal pathologies presenting as acute abdomen have not been described in any previous study in terms of presentation, management and outcome.

Objectives: The objective of this study was to identify the reported causes of primary cecal pathologies presenting as acute abdomen and the various causes presenting in Indian setting, to discuss morbidity and mortality associated with cecal pathologies and to critically analyse the various management modalities employed in emergency setting.

DETAILED DESCRIPTION:
The importance of cecal pathologies lie in the fact that being the first part of large intestine, any disease involving the cecum affects overall functioning of the large bowel. Primary cecal pathologies presenting as acute abdomen often pose a challenge to their optimal management due to requirement of urgent intervention in most cases and being a common source of misdiagnosis. These pathologies often mimic acute appendicitis and commonly misdiagnosed as one. This misdiagnosis can lead to under-treatment of the underlying pathology and this results in high morbidity and mortality associated with these conditions. So the accurate identification of such conditions is required so that the patients can be optimally managed and patient outcome can be improved.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients presenting in emergency department with acute abdomen were included in study in whom cecal pathology as the cause of acute abdomen was suspected clinically and/or on imaging and further confirmed per-operatively and/or on histopathological examination (HPE) or on imaging. Patients identified with primarily a cecal pathology who had acute pain abdomen as the initial symptom but who didn't presented immediately due to various reasons were also included in the study as it is a well-documented fact that patients in developing countries like India, especially those who live in rural areas or who are illiterate often resort to indigenous methods of treatment or take symptomatic treatment from local practitioners before presenting to a tertiary centre for definitive treatment. Also, only those patients who were operated within 24 hours of index admission in the emergency operation theatre (EOT) by a registrar or faculty member after initial resuscitation were included in the study.

Exclusion Criteria:

* Patients with sub-acute, intermittent or chronic pain; when predominant symptoms were attributable to some other cause even with concomitant presence of a cecal pathology; when predominant pathology was not cecal and patients with cecal pathology operated as an elective case were excluded from this study. Thus patients diagnosed to be having appendiceal stump blowout, perforation of base of appendix, ileocecal tuberculosis or intussusception were not included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients presenting in the emergency department with acute abdomen were included in study in whom cecal pathology as the cause of acute abdomen was suspected clinically and/or on imaging and further confirmed per-operatively and/or on histopathological examination (HPE) or on imaging.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-07-15 (Actual)

PRIMARY OUTCOMES:
Pattern of primary cecal pathology in Indian setting | 10 years
  The objective of this study was to identify the reported causes of cecal pathology presenting as acute abdomen in medical literature and the various causes presenting in Indian setting, to identify the pattern of common pathologies in Indian setup, to discuss morbidity and mortality associated with cecal pathologies and to critically analyse the various management modalities commonly employed for cecal pathologies presenting as acute abdomen.

CONTACTS AND LOCATIONS:
Overall Officials: Kaushal D Singh, MS Surgery, Principal Investigator — Jawaharlal Nehru Medical College, Aligarh

IPD SHARING:
Plan to Share IPD: Undecided
Data can be shared on request for multi-institutional prospective studies.

DOCUMENTS (2):
  • Study Protocol (2016-01-01): https://cdn.clinicaltrials.gov/large-docs/25/NCT03262025/Prot_000.pdf
  • Informed Consent Form (2016-01-01): https://cdn.clinicaltrials.gov/large-docs/25/NCT03262025/ICF_001.pdf